CLINICAL TRIAL: NCT03950024
Title: Contribution of Functional Brain MRI to the Understanding of Arthrogenic Muscle Inhibition (AMI) in the Aftermath of Knee Trauma.
Brief Title: Improvement of Knowledge About the Arthrogenic Muscle Inhibition in the Aftermath of Knee Trauma.
Acronym: CAMIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/19/0029; 2019-A00479-48 (Other: ANSM)
Record Dates: First submitted 2019-05-09; First posted 2019-05-14 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: arthrogenic muscle inhibition; anterior cruciate ligament; functional brain MRI; Central nervous system; Knee trauma
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: prospective, monocentric, interventional, comparative, controlled, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with arthrogenic Muscle Inhibition (Experimental)
  Interventions: Diagnostic Test: functional brain MRI
- without arthrogenic Muscle Inhibition (Active Comparator)
  Interventions: Diagnostic Test: functional brain MRI

INTERVENTIONS:
Diagnostic Test: functional brain MRI — The functional brain MRI realized will be a examination with a resting sequence and a sequence during a movement imagination task. (knee bent)

SUMMARY:
Arthrogenic Muscle Inhibition (AMI) is one of the classic complications occurring in the aftermath of knee trauma; AMI is grossly defined as a lack of extension due to quadriceps inhibition and hamstring contracture. However, its origins remains unknown with a strong suspicion for a central brain origin. It could be the missing link explaining this lack of extension following an anterior cruciate ligament (ACL) rupture. The primary hypothesis of this study is that a difference in activation of motor brain areas exists in patients with an ACL rupture, between those with AMI or without. The second hypothesis is that this difference could be seen on brain functional MRI.

DETAILED DESCRIPTION:
AMI leads to quadriceps atrophy, persistent knee pain, dynamic instability, and a higher rate of osteoarthritis. A recent literature review suggests that the AMI phenomenon is multifactorial, but not widely known and poorly understood. Known mechanisms include impaired motor function at rest, impaired transmission of information from joint sensory receptors, impaired excitability of the spinal reflex and impaired cortical activity. Several studies have suggested a link between ACL rupture and central nervous system reorganization. Among the neurophysiological investigations explored are the evoked somesthesic potentials, electroencephalography, and transcranial magnetic stimulation (TMS). However, these mechanisms alone do not explain the phenomenon in its entirety, suggesting that there are other mechanisms. Furthermore, no study has used functional brain MRI to assess the existence of similar changes in AMI.

This study plans to compare two groups of patients with an ACL rupture: a group with AMI, and a group without AMI. Both groups will undergo a functional brain MRI in order to analyse any modification of the sensory-motor network connectivity that could occur.

ELIGIBILITY:
Inclusion Criteria:

* male patient, right-handed,
* with a severe right knee sprain in the event of ACL rupture,
* occurrence of trauma within 4 weeks prior to inclusion,
* with a score of ≥ 8/10 on the Edinburgh Manual Laterality Questionnaire, -affiliated or benefiting from public health services.

Exclusion Criteria:

* person presenting any of these conditions : professional player / athlete, -contraindication to the MRI examination (claustrophobic patient, patient with a metallic element),
* patient already operated on with ligament damage to the knee other than ACL,
* patient with iterative ACL rupture,
* patient who has undergone contralateral ligament reconstruction,
* patient with multi-ligamentary knee injury,
* patient refusing to be informed of any abnormality detected on brain MRI, -protected patient (adults under guardianship or other legal protection, deprived of their liberty by judicial or administrative decision).

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Matrix of correlation coefficients | Day 0
  A matrix of correlation coefficients, measured by MRI, representing the strength of the sensory-motor network connectivity at rest for each group.

SECONDARY OUTCOMES:
Activation map of the motor representations of knee movement | Day 0
  An activation map of the motor representations of knee movement are measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Etienne CAVAIGNAC, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Pierre Paul Riquet Hospital, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No